CLINICAL TRIAL: NCT01507038
Title: Phase II Clinical Trial to Investigate the Efficacy, Safety and Pharmacokinetics of YH14617 After Once Weekly or Biweekly Administration in Patients With Type 2 Diabetes Mellitus
Brief Title: Safety and Efficacy of YH14617 in Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Collaborators: Peptron, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YH14617-201
Record Dates: First submitted 2012-01-05; First posted 2012-01-10 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; YH14617; Exenatide; Yuhan
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group A (Experimental)
  Interventions: Drug: YH14617
- Group B (Experimental)
  Interventions: Drug: YH14617
- Group C (Experimental)
  Interventions: Drug: YH14617
- Group D (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: YH14617 — 1mg once weekly
  Arms: Group A
Drug: YH14617 — 1.6mg once weekly
  Arms: Group B
Drug: YH14617 — 2mg once biweekly
  Arms: Group C
Drug: Placebo — Once weekly
  Arms: Group D

SUMMARY:
The objective of this study is to assess the safety, efficacy and pharmacokinetic of YH14617 after once weekly or biweekly injection in patients with type 2 Diabetes Mellitus to investigate the optimal recommended dosage. Study period is 20 weeks including 12 weeks of treatment period and 8weeks of follow-up period without treatment.

ELIGIBILITY:
Inclusion Criteria:

* Have signed a written informed consent voluntary, prior to the any procedure
* Volunteers of aged between 20 years to 75 years
* Have been diagnosed with type 2 diabetes at least 3 months prior to study
* Have a body mass index (BMI) of > 23kg/m2 and have a history of stable body weight during 3 months prior to the first administration (not varying by > 5% in weight)
* Have been treated with stable dose regimen of Metformin > 1500mg/day or maximum tolerant dose for at least 3 months prior to the first administration
* Have an HbA1c between 7% and 10% inclusive

Exclusion Criteria:

* Have been treated with insulin, sulfonylurea, thiazolidinedione class hypoglycemic drugs, exenatide or other GLP-1 receptor agonist, DPP4-inhibitor, glucocorticoid and drugs that promote weight loss within 3 months prior to the first administration
* Have acute disease, other untreated disease or diabetic complications that needs additional treatment
* Have severe renal disorder(serum creatinine concentration > 1.5 times of normal upper limit) or liver disorder(liver enzyme > 2 times of normal upper limit)
* Have blood pressure > 160/100mmHg
* Have been hospitalized due to cardiac disorder(angina, cardiac infarction, heart failure and etc.) within 1 year prior to the first administration
* Have history of critical disease within 1 year prior to the first administration
* Have untreated malignant tumor or have history of significant malignant tumor within 5 years prior to the first administration
* Have fasting plasma glucose(FPG) > 250mg/dl or have random glucose level > 350mg/dl
* Have more than 1 history of severe hypoglycemia that needed others help within 3 months prior to the first administration
* Have a known allergy or hypersensitivity to drugs
* Pregnant women, nursing mothers or subject who does not agree to assigned contraception in the study
* Participated in any other clinical trials within 30 days prior to the first administration
* Subject who is judged to be ineligible by principal investigator or sub-investigator according to various reasons other than above

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2011-12; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c at week 12 | Baseline, Week 12

SECONDARY OUTCOMES:
Change from baseline in body weight at week 12 | Baseline, Week 12
Change from baseline in fasting plasma glucose at week 12 | Baseline, Week 12
Change from baseline in 1,5-anhydroglucitol at week 12 | Baseline, Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Seop Choi, MD, PhD., Principal Investigator — Korea University Anam Hospital
Locations (1):
- Yuhan, Seoul, South Korea